CLINICAL TRIAL: NCT02351531
Title: Cow Milk Allergy: Evaluation of the Efficacy of a New Thickened Extensively Hydrolyzed Formula in Infants With Confirmed Cow Milk Allergy
Acronym: COMETE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UP-2013-02
Record Dates: First submitted 2015-01-21; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Cow Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- New Thickened Extensively Hydrolyzed formula (Experimental)
  Interventions: Dietary Supplement: Extensively Hydrolyzed formula

INTERVENTIONS:
Dietary Supplement: Extensively Hydrolyzed formula

SUMMARY:
The aim of the study is to assess the hypoallergenicity of a new thickened extensively hydrolyzed formula.

ELIGIBILITY:
Inclusion Criteria:

* between 1 and 12 months old
* having a cow milk allergy confirmed by a positive double-blind food challenge performed in the last 3 months,
* whose parent(s) signed the informed consent form

Exclusion Criteria:

* Infants mainly or exclusively breastfed,
* Infants having a weight at inclusion < 2500g,
* Infants who refused to drink an extensively hydrolyzed formula anytime prior to inclusion,
* Infants fed an amino acid based formula
* Infants who had an anaphylactic reaction in the past,

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of patients dropped out for intolerance | 2 weeks

SECONDARY OUTCOMES:
Cow's milk protein hypersensitivity score | 2 weeks
Growth (weight, height, head circumference) | 3 months
Growth (weight, height, head circumference) | 4 months

CONTACTS AND LOCATIONS:
Locations (3):
- Centre Hospitalier Régional, Namur, Belgium
- Necker Children's Hospital, Paris, France
- University of Naples Federico II, Naples, Italy

REFERENCES:
- [Derived] Dupont C, Bradatan E, Soulaines P, Nocerino R, Berni-Canani R. Tolerance and growth in children with cow's milk allergy fed a thickened extensively hydrolyzed casein-based formula. BMC Pediatr. 2016 Jul 18;16:96. doi: 10.1186/s12887-016-0637-3. PMID 27430981